CLINICAL TRIAL: NCT03496402
Title: Molecular and Immunological Characterisation of High Risk CHildhood Cancer At DiagnOsis, Treatment and Follow-up - Biological Evaluation in Children, Adolescents and Young Adults -
Brief Title: Biological Characterisation of High Risk CHildhood Cancer in Children, Adolescents and Young Adults (MICCHADO)
Acronym: MICCHADO
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Institut Curie (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: IC 2017-02
Record Dates: First submitted 2018-02-26; First posted 2018-04-12 (Actual); Last update posted 2025-03-18 (Actual); Status verified 2025-03

CONDITIONS: Neuroblastoma; Rhabdomyosarcoma; Ewing Sarcoma Family of Tumors; Osteosarcoma; Leukemia; Central Nervous System Tumor
MeSH Terms: conditions — Neuroblastoma; Rhabdomyosarcoma; Neuroectodermal Tumors, Primitive, Peripheral; Osteosarcoma; Leukemia; Central Nervous System Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- High risk Cohorts (Experimental): Cohort 1 : High risk Neuroblastoma, High risk Rhabdomyosarcoma, High risk Ewing Sarcoma Family Tumor, High risk Osteosarcoma, High risk Leukaemia (secondary acute myeloid leukaemia or biphenotypic acute leukaemia) Cohort 2 : Extracerebral and cerebral high risk tumor, High risk Leukaemia (leukaemia with high MRD) Sampling on blood, bone marrow and cerebrospinal fluid
  Interventions: Other: Sampling on blood, bone marrow and cerebrospinal fluid
- Low risk Cohort (Experimental): Cohort 3 : Intermediate or low risk tumors : Neuroblastoma, Rhabdomyosarcoma, Ewing Sarcoma Family Tumor, Osteosarcoma Sampling on blood, bone marrow and cerebrospinal fluid
  Interventions: Other: Sampling on blood, bone marrow and cerebrospinal fluid

INTERVENTIONS:
Other: Sampling on blood, bone marrow and cerebrospinal fluid — biological sampling during treatment and follow-up

SUMMARY:
Methodology:

Prospective, multicentric, open, non-randomised, non-therapeutic, interventional study

DETAILED DESCRIPTION:
To identify and characterise:

* meaningful molecular genetic alterations,
* meaningful immunological features of high risk childhood, adolescents and young adult cancers, at diagnosis, during patient treatment and follow-up (time dimension).

ELIGIBILITY:
Inclusion Criteria:

1. Inclusion within 3 months after diagnosis
2. Availability of a cryopreserved tumour sample (primary and/or metastatic and/or lymph nodes) or peripheral blood or bone marrow samples (if invasion more than 30% of lymphoblasts) for leukaemias, obtained at the time of diagnosis during a routine procedure
3. Availability of a formalin-fixed paraffin-embedded (FFPE) tumour sample (primary and/or metastasis and/or lymph nodes), obtained at the time of diagnosis during a routine procedure (except for leukaemia patients)
4. Age: ≤ 25 years at diagnosis
5. Written patient informed consent, or parents or legal representative written informed consent and assent of the child and the adolescent
6. Compulsory affiliation to a social security scheme

   Additional inclusion criteria for the study:

   To avoid multiple sampling for children, adolescents and young adults with cancer, patients already included or to be included in a study with similar analyses and/or objectives might also be included in MICCHADO study and in this case, samples or data might be exchanged on a collaborative basis.

   Cohort 1:
   * High risk neuroblastoma:

     - Any type of neuroblastoma with MYCN amplification, except INSS stage 1

     - Stage 4 neuroblastoma in children older than one year at diagnosis
   * High risk rhabdomyosarcoma:

     * Foxo1 rearrangement any stage;
     * and / or N1 ;
     * and / or metastatic rhabdomyosarcoma
   * High risk Ewing sarcoma:

     * Metastatic Ewing sarcoma family of tumours (ESFT)
     * Localised inoperable Ewing sarcoma with primary tumours ≥ 200 ml
   * High risk osteosarcoma:

     - Metastatic osteosarcoma

     - Localised inoperable osteosarcoma
   * High risk leukaemia:

     * Secondary acute myeloid leukaemia
     * Biphenotypic acute leukaemia

   Cohort 2:

   • Extra cerebral or cerebral high risk tumours including:
   * other metastatic sarcomas,
   * other rare high risk cancers,
   * high risk renal tumours with surgery after an initial chemotherapy
   * rhabdoid brain tumours (AT/RT) and extra cerebral rhabdoid tumours
   * high risk or metastatic cancers of unclear histological diagnosis • Lymphoblastic leukaemia with high MRD at Day 78 (time point 2) • Very high risk T-cells acute lymphoblastic leukaemia:
   * MRD ≥ 10-2 at the end of the induction ;
   * or MRD ≥ 10-3 at Day 78

   Cohort 3:

   Children, adolescents and young adults, with low/intermediate risk cancers belonging to the following types:

   • Neuroblastoma:

   - Localised, without MYCN amplification
   * Localised, INSS stage 1, with MYCN amplification
   * Stage 4s, in infants (younger than one year at diagnosis), without MYCN amplification

     • Rhabdomyosarcoma:
   * Localised, without Foxo1 rearrangement

     • ESFT:
   * All non-high risk localised ESFT • Osteosarcoma:
   * All non-high risk localised osteosarcoma

   Exclusion Criteria:

   Main non-inclusion Criteria common to all study cohorts:

1) Age: patients > 25 years old at diagnosis 2) Absence of patient or parents or legal representative written informed consent 3) Patient for whom follow-up by the investigating centre does not appear feasible

Ages: 1 Year to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 600 (Estimated)
Dates: Start 2018-04-20 (Actual); Primary Completion 2027-04-19 (Estimated); Study Completion 2027-08-19 (Estimated)

PRIMARY OUTCOMES:
Number of patients with meaningful molecular genetic alterations | At the end of study (6 years)
  Identification of molecular genetic alterations based on molecular characterisation of tumor at diagnosis, during patient treatment and follow-up (time dimension)
Number of patients with meaningful immunological features | At the end of study (6 years)
  Identification and characterisation of the tumor microenvironment and the host's immunological profile, at diagnosis and during patient treatment
Number of patients with identification of new tumor-specific genetic characteristics during follow-up (clonal evolution) | up to 6 years
  Comparison between genetic variations identified at diagnosis and those identified on circulating tumor DNA during treatment, FU and/or relapse

SECONDARY OUTCOMES:
Correlation between disease recurrence and molecular and/or immunological biomarkers | up to 6 years
  To characterise biomarkers, based on molecular analyses of tumour samples from diagnosis, for prognostic and predictive purposes.
  To characterise the tumour microenvironment and the host's immunological profile, for prognostic and predictive purposes.
  To identify potential prognostic and predictive biomarkers on samples collected during patient's treatment and follow-up, based on changes on circulating tumour DNA (ctDNA), detected by molecular biology techniques, and on immunological findings
Correlation between genetic variations and immune parameters | up to 6 years
  To compare molecular and immunological findings at diagnosis and during treatment (data integration)
Correlation between disease staging and immunological features | up to 6 years
  To investigate the impact of the tumour microenvironment and host's immunological profile on the disease staging at diagnosis, by comparing patients with metastatic to patients with localised disease

CONTACTS AND LOCATIONS:
Overall Officials: Gudrun SCHLEIERMACHER, MD, Principal Investigator — Institut Curie
Locations (30):
- France (30):
  - Chu D'Amiens Picardie, Amiens
  - CHU Angers, Angers
  - CHRU de Besançon - Hôpital Jean-Minjoz, Besançon
  - CHU de Bordeaux - Hôpital des enfants - Groupe Hospitalier Pellegrin, Bordeaux
  - CHRU de Brest, Brest
  - CHU CAEN, Caen
  - Centre Régional de Cancérologie et Thrapie Cellulaire Pdiatrique (CRCTCP), Clermont-Ferrand
  - CHU Hôpital d'Enfants, Dijon
  - CHU GRENOBLE Alpes - Hôpital Couple-Enfant, Grenoble
  - Centre Oscar Lambret, Lille
  - CHU de Limoges - Hôpital Mère-Enfant, Limoges
  - Centre Léon Bérard, Lyon
  - Hospices Civils de Lyon, Lyon
  - Hôpital d'Enfants de la Timone (AP-HM), Marseille
  - CHU Arnaud de Villeneuve, Montpellier
  - CHU Nantes - Hôpital Mère Enfant, Nantes
  - Hôpital l'Archet 2, Nice
  - Hôpital d'Enfants Armand-Trousseau, Paris
  - Hôpital universitaire Robert-Debré (AP-HP), Paris
  - Institut Curie, Paris
  - CHU de Poitiers, Poitiers
  - CHU de Reims - Hôpital Américain, Reims
  - Chu Hopital Sud Rennes, Rennes
  - CHU de Rouen - Hôp. Charles NICOLLE, Rouen
  - CHU Saint-Etienne - Hôpital Nord, Saint-Etienne
  - Hôpitaux Universitaires de Strasbourg - Hôpital de Hautepierre, Strasbourg
  - CHU Hôpital des Enfants, Toulouse
  - CHU TOURS - Hôpital Clocheville, Tours
  - CHU Nancy - Hôpital d'Enfants, Vandœuvre-lès-Nancy
  - Gustave Roussy, Villejuif

IPD SHARING:
Plan to Share IPD: No